CLINICAL TRIAL: NCT02641613
Title: The Efficacy of Retroclavicular Versus Supraclavicular Brachial Plexus Block in Patients Undergoing Forearm and Hand Surgery: a Randomized Controlled Double-blinded Trial.
Brief Title: Retroclavicular Versus Supraclavicular Brachial Plexus Block for Hand and Forearm Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hôpital du Valais (Other)
Responsible Party: Principal Investigator, Sina Grape, MD, Hôpital du Valais
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCVEM 038/15
Record Dates: First submitted 2015-12-01; First posted 2015-12-29 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Hand Injury
MeSH Terms: conditions — Hand Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- supraclavicular (Active Comparator): patients receive a supraclavicular block for forearm or hand surgery with 30 ml of a mixture of ropivacaine 0.5 % and mepivacaine 1 %
  Interventions: Procedure: supraclavicular block
- retroclavicular block (Experimental): patients receive a retroclavicular block for forearm or hand surgery with 30 ml of a mixture of ropivacaine 0.5 % and mepivacaine 1 %
  Interventions: Procedure: retroclavicular block

INTERVENTIONS:
Procedure: retroclavicular block — retroclavicular block for forearm or hand surgery
  Arms: retroclavicular block
Procedure: supraclavicular block — supraclavicular block for forearm or hand surgery
  Arms: supraclavicular

SUMMARY:
Patients will be randomized to one of two groups:

1. Supraclavicular group: supraclavicular brachial plexus block performed with the aid of ultrasound;
2. Retroclavicular group: retroclavicular brachial plexus block performed with the aid of ultrasound.

DETAILED DESCRIPTION:
The study will be proposed to all patients undergoing formarm or hand surgery under brachial plexus block. Patients will be randomized to one of two groups The first group - supraclavicular group - will receive an ultrasound-guided brachial plexus block via the supraclavicular approach, by injection of 30 ml of a mixture of ropivacaine 0.5 % + mepivacaine 1 %. The second group - retroclavicular group - will receive an ultrasound-guided brachial plexus block via the retroclavicular approach, by injection of 30 ml of a mixture of ropivacaine 0.5 % + mepivacaine 1 %. Primary outcome is success rate at 30 minutes after the injection defined as loss of sensation to pinprick in the forearm and hand. Secondary outcomes are: needling time, time to first analgesic request, postoperative opioid consumption, pain scores at 12 and 24 hours postoperatively, block-related complications, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who undergo forearm or hand surgery under brachial plexus block.

Exclusion Criteria:

* History of allergic reaction to local anaesthetics

  * Peripheral neuropathy
  * Renal or hepatic insufficiency
  * Coagulation disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-01; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Success rate (loss of sensation to pinprick in the forearm and hand) | 30 minutes after the injection

SECONDARY OUTCOMES:
Needling time in seconds | 15 min
Time to first analgesic request | 24 hours
Block-related complications | 24 hours
Postoperative opioid consumption on postoperative day 1 | 24 hours
Pain scores at 12 hours postoperatively | 12 hours
  measured on a visual analogue scale between 0 and 100
Pain scores on postoperative day 1 | 24 hours
  measured on a visual analogue scale between 0 and 100
Patient satisfaction as assessed by numerical rating scale | 24 hours
  Patient satisfaction on a scale between 0 (= completely dissatisfied) and 10 (= completely satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Sina Grape, MD, Principal Investigator — Hopital du Valais; Eric Albrecht, MD, Study Director — CHUV
Locations (1):
- Hopital du Valais, Sion, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Grape S, Pawa A, Weber E, Albrecht E. Retroclavicular vs supraclavicular brachial plexus block for distal upper limb surgery: a randomised, controlled, single-blinded trial. Br J Anaesth. 2019 Apr;122(4):518-524. doi: 10.1016/j.bja.2018.12.022. Epub 2019 Jan 31. PMID 30857608